CLINICAL TRIAL: NCT06255873
Title: Effects of L-Carnitine Supplementation on Gastric Emptying in Children With Drug Resistant Epilepsy on Ketogenic Diet
Brief Title: Effects of L-Carnitine on Gastric Emptying in Children With Drug Resistant Epilepsy on Ketogenic Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 630/ 2022
Record Dates: First submitted 2024-02-03; First posted 2024-02-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ketogenic Diet
MeSH Terms: interventions — Carnitine; Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketogenic diet with L - Carnitine supplementation. (Experimental): Patients with drug resistant epilepsy who received ketogenic diet with L - Carnitine supplementation.
  Interventions: Dietary Supplement: L- Carnitine; Other: ketogenic diet
- ketogenic diet. (Active Comparator): Patients with drug resistant epilepsy who received ketogenic diet only.
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Dietary Supplement: L- Carnitine — L-carnitine was taken after feeds in the form of tablets or dissolved tablets in a dose of 50 mg/kg/day, with maximum dose of 2 g/day.
  Arms: ketogenic diet with L - Carnitine supplementation.
Other: ketogenic diet — ketogenic diet (KD) initiated under supervision of expert physician who considered patient's age, type of feeding, needs and preferences of the child and his/her family to select the type and initial ratio of KD therapy, KD ratio ranged from 1:1 to 4:1 of lipids to carbohydrates plus proteins in grams.

SUMMARY:
This study was conducted on thirty children aged from12 months to 18 years newly diagnosed with drug resistant epilepsy and following up at Pediatric Nutrition and Neurology Outpatient Clinics assigned randomly into 2 groups, group1: patients who started ketogenic diet with L-carnitine and group2: patients who started ketogenic diet only.

ELIGIBILITY:
Inclusion Criteria:

* All infants and children aged from 12 months to 18 years old newly diagnosed with drug resistant epilepsy and were assigned to start KD.

Exclusion Criteria:

* Patients with intolerance or non-compliance to ketogenic diet therapy.
* Patients for epilepsy surgery or vagal nerve stimulation.
* Children with history of previous abdominal operations.
* Children with history of GI diseases affecting GI motility before starting KD.
* Children with tube feeding or feeding gastrostomy or jejunostomy.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Assessment the effect of L-carnitine supplementation on gastric emptying in children with drug resistant epilepsy (DRE) on ketogenic diet (KD). | At time of enrollment and 3 months of intervention.
  Antral length measurement using abdominal ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: May F Nassar, MD, Study Director — Professor of pediatrics, Faculty of Medicine, Ain shams University
Locations (1):
- Faculty of Medicine-Ain Shams University, Cairo, Abbasia, Egypt